CLINICAL TRIAL: NCT06127979
Title: Differential Changes in Ki67 Between Carriers and Noncarriers of BRCA2 Mutations With Estrogen Receptor-Positive, Human Epidermal Growth Factor Receptor 2-negative Breast Cancer Treated With Preoperative Endocrine Therapy
Brief Title: A Study of Changes in Ki67 Expression in People With Breast Cancer Receiving Endocrine Therapy Before Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 23-311
Record Dates: First submitted 2023-11-06; First posted 2023-11-13 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Breast Cancer
Keywords: Ki67 Expression; BRCA2 mutation; ER+/HER2-; endocrine therapy; 23-311
MeSH Terms: conditions — Breast Neoplasms | interventions — Biopsy, Large-Core Needle; Blood Specimen Collection

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Breast Cancer (Experimental): All study patients will receive standard ET for at least 2 weeks. In accordance with the standard of care, postmenopausal women will receive AI (anastrazole 1mg daily tablet, letrozole 2.5mg daily tablet, or exemestane 25mg daily tablet Which will be followed by standard of care surgical treatment. Surgical tumor tissue will be obtained at the time of surgery and will be assessed for Ki67; a portion of this specimen will be snap-frozen for future analysis. In collaboration with the surgical team, Oncotype can be sent on this research biopsy after pathology assessment. This will enable the patient to receive the Oncotype result and to gain knowledge on the recommendation for adjuvant chemotherapy about 4-6 weeks earlier than our normal workflow.
  Interventions: Procedure: core needle biopsy; Other: blood draw

INTERVENTIONS:
Procedure: core needle biopsy — Pre-Endocrine Therapy core needle biopsy. The pre-treatment research biopsy will require a biopsy marker clip to document that the cancer lesion was biopsied
Other: blood draw — blood draw

SUMMARY:
The researchers are doing this study to look at changes in Ki67 expression after at least 2 weeks of endocrine therapy in people with ER+/HER2- breast cancer undergoing cancer removal surgery. Participants will receive the endocrine therapy before their surgery. The researchers will look at how changes in Ki67 expression compare between participants who are carriers of the BRCA2 mutation and participants who are noncarriers of the BRCA2 mutation.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women aged ≥18 years with biopsy-proven stage I-III invasive breast cancer that is ER+/HER2-
* Scheduled to undergo upfront surgery
* Eligible for genetic testing in accordance with National Comprehensive Cancer Network guidelines(BRCA2 arm only)

Exclusion Criteria:

* History of breast cancer
* Receipt of ET for risk reduction in the previous 3 months
* Stage IV disease at presentation
* Scheduled to undergo neoadjuvant systemic chemotherapy
* Pregnant

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Breast Cancer
Enrollment: 42 (Estimated)
Dates: Start 2023-11-06 (Actual); Primary Completion 2028-11 (Estimated); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
assess the change in Ki67 | baseline to at least 2 weeks of endocrine therapy
  The change in Ki67 expression on immunohistochemical staining from baseline to at least 2 weeks of ET will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Minna Lee, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center (All Protocol Activities), New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm